CLINICAL TRIAL: NCT06914843
Title: A Randomized Controlled Pilot of a Web-based Intervention for Cognitive Behavioral Therapy-based Training to Improve Mental Health in Medical Trainees
Brief Title: Digital Intervention to Promote Medical Trainee Well-being (OptimalWork Pilot)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Ginger E Nicol, Associate Professor of Psychiatry (Child), Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 202208152
Record Dates: First submitted 2024-07-24; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2024-12

CONDITIONS: Mental Health Wellness 1
Keywords: Cognitive Behavioral Therapy; Digital Mental Health

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants are randomized using a digital data management platform (REDCap) and investigators and analysts remain blinded to participant identifiers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OptimalWork (Experimental): An online intervention that teaches concepts of cognitive restructuring, mindfulness, and behavioral activation as they apply in one's daily life and work. Users are given personalized content recommendations based on their inventory results and instructed to complete 15-25 minutes of content per day, 5 days/week for 4 weeks.
  Interventions: Behavioral: OptimalWork
- Podcast Listening (Active Comparator): A curated series of podcasts on topics unrelated to cognitive behavioral therapy or mindfulness, modeled after a similar control from a study of a mindfulness based intervention (Basso et al. 2019). Users are instructed to complete one podcast per day on a digital platform (~15 minutes/day), 5 days/week for 4 weeks.
  Interventions: Behavioral: Podcast Listening

INTERVENTIONS:
Behavioral: OptimalWork — An online intervention that teaches concepts of cognitive restructuring, mindfulness, and behavioral activation as they apply in one's daily life and work. Users are given personalized content recommendations based on their inventory results and instructed to complete 15-25 minutes of content per day, 5 days/week for 4 weeks. (optimalwork.com)
  Arms: OptimalWork
Behavioral: Podcast Listening — A curated series of podcasts on topics unrelated to cognitive behavioral therapy or mindfulness, modeled after a similar control from a study of a mindfulness based intervention (Basso et al. 2019). Users are instructed to complete one podcast per day on a digital platform (~15 minutes/day), 5 days/week for 4 weeks.
  Arms: Podcast Listening

SUMMARY:
This project aims to address stress, anxiety, burnout, and depression among medical trainees using a web-based intervention that teaches cognitive behavioral therapy (CBT)-based skills to increase resilience. The intervention is a web application ("OptimalWork", optimalwork.com) that includes a "MasterClass" consisting of about 20 interactive modules to be completed over four weeks (five days/week, 15-25 minutes/day). These modules teach principles and skills of CBT in an interactive manner and give tailored recommendations for how to apply and develop these skills in one's work and personal life. Participants who enroll in the study will be randomly assigned to either the MasterClass intervention or an active control (podcast listening) condition, and the control group will be given access to the MasterClass after 8 weeks. Measurements of well-being at baseline, 4 weeks, 8 weeks, 12 weeks, and 16 weeks will be compared between the groups as the primary outcome. Participant engagement as measured by MasterClass module completion and qualitative feedback will also be collected to guide future efforts at large-scale implementation in medical trainees and healthcare workers.

DETAILED DESCRIPTION:
Medical students face significant mental health challenges, with burnout being a prevalent concern. Given the efficacy of cognitive behavioral therapy (CBT) and mindfulness-based approaches for treating mood and anxiety disorders, many individual-level interventions to reduce stress or prevent burnout have focused on teaching people these psychological skills, including digital approaches that aim to overcome the barriers to implementation of face-to-face therapy.

One such digital intervention is OptimalWork (optimalwork.com), an online platform that teaches CBT- and mindfulness-based skills as they apply in daily life and work. The focus of the intervention is learning to reframe challenges in one's everyday work as opportunities to grow according to one's ideals and to strengthen one's bonds with others. Our primary aims are to determine the feasibility, acceptability, and preliminary effect size of this intervention in medical students. We also aim to describe relationships between different measures of well-being, including some that measure clinical symptoms and others that measure flourishing. Finally, we aim to identify barriers and facilitators to successful implementation in this population through exit interviews and other qualitative feedback.

We are conducting a 16-week randomized controlled trial, comparing the OptimalWork online program versus a Podcast Listening control group (described below). Podcasts were chosen from RadioLab to last about the same time as the OptimalWork program (10-15 minutes / day, 5 days / week for 4 weeks) but with content unrelated to wellness or mental health. The intervention period lasts 4 weeks, and outcome measures (surveys) are administered at baseline, 4, 8, 12, and 16 weeks. After 8 weeks and completion of the second follow-up survey, participants are given the option to access the other intervention if they so desired. This is to ensure equity in access to the intervention between groups.

Eligible participants are students currently enrolled at Washington University School of Medicine from all class years (M1-M4, including those on research years and MD/PhD students in the PhD years). Participants must not be participating in another behavioral health or well-being intervention at the time of enrollment. We are not excluding participants based on mental health diagnosis or active treatment.

All participants provide informed consent electronically after reviewing the nature, risks, and benefits of the study, under protocols approved by the Washington University Human Research Protection Office.

Our primary outcomes at 8 weeks are: (1) Flourishing as assessed by the Human Flourishing Index (HFI) a broad, well-validated measure based around five domains (Happiness and Life Satisfaction, Mental and Physical Health, Meaning and Purpose, Character and Virtue, and Close Social Relationships); (2) Work engagement as assessed by the OptimalWork Inventory (OWI), comprised of four sub-domains (Friendships, Ideals, Mode of Working, Work-Life Harmony); and (3) Burnout as measured by the Professional Fulfillment Index (PFI), particularly the two domains of Interpersonal Disengagement and Work Exhaustion.

Secondary outcomes assess four additional domains: (1) Emotional Support (Patient-Reported Outcomes Measurement Information System ("PROMIS") - Emotional Support, 4 items); (2) Anxiety (PROMIS - Anxiety, 4 items); (3) Depression (PROMIS - Depression, 4 items); and (4) Stress (Brief Inventory of Perceived Stress, BIPS). The Stress measure comprises three sub-domains: Pushed, Conflict and Imposition, and Lack of Control. These measures are all reported on a 5-point Likert Scale. We also include a one-item sleep assessment (Sleep Quality Scale, self-rated from 1-10).

For statistical analyses, we will use repeated-measures mixed models to look at trajectories over 4 and 8 weeks with a time*intervention group interaction term to estimate the effect of the OptimalWork intervention on these well-being domains over time. Longer-term effects of the intervention on well-being measurements at 12- and 16-week follow-up were also assessed with similar models. Secondary analyses included between-group comparisons of trajectories of sub-domains of HFI, OWI, and PFI, as well as secondary outcomes (Emotional Support, Anxiety, Depression, Stress), modeled as above.

If successful, our findings will have implications for the feasibility, acceptability, and effectiveness of these sorts of interventions, with the long-term goal of informing future interventions targeting medical student well-being.

ELIGIBILITY:
Inclusion Criteria:

* Current or incoming WashU School of Medicine Student

Exclusion Criteria:

* Currently participating in another behavioral health / well-being intervention
* Unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-09-06 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Human Flourishing Index | 8 weeks
  Broad well-being based around 5 domains of happiness, mental and physical health, meaning and purpose, character and virtue, and close social relationships.
OptimalWork Inventory | 8 weeks
  24-item survey designed to measure how well one is engaging challenges in one's work and personal life

SECONDARY OUTCOMES:
Stress - BIPS | 8 weeks
  Brief Inventory of Perceived Stress
Burnout and professional fulfillment | 8 weeks
  Professional Fulfillment Index (7 items)
Anxiety - PROMIS | 8 weeks
  4-item survey from the Patient Reported Outcomes Measurement Information System
Depression - PROMIS | 8 weeks
  4-item depression inventory from the Patient-Reported Outcomes Measurement Information System

CONTACTS AND LOCATIONS:
Overall Officials: Ginger E. Nicol, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanchez JS, Perry D, Kinghorn A, Vermette D, Gray T, Duncan JG, Evanoff B, Nicol GE. Optimizing the Work of Learning for Flourishing: A Randomized Pilot Study of a Digital CBT-Based Intervention in Medical Students. Acad Psychiatry. 2026 Feb 7. doi: 10.1007/s40596-026-02308-w. Online ahead of print. PMID 41652149